CLINICAL TRIAL: NCT01871597
Title: Ex-Vivo Evaluation of the Effectiveness of Pulmonary Artery Sealing for VATS Procedure
Brief Title: Pulmonary Artery Energy Sealing for VATS Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0041
Record Dates: First submitted 2013-05-14; First posted 2013-06-07 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Lung Cancer
Keywords: Lung cancer; VATS procedure; Pulmonary Artery Sealing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Group (Experimental): Intervention - Pulmonary Artery Energy Seal
  Interventions: Device: Pulmonary Artery Energy Seal

INTERVENTIONS:
Device: Pulmonary Artery Energy Seal — Pulmonary artery energy seal devices such as: Ligasure, Harmonic scalpel, Enseal, Thunderbeat, Unipolar and Conventional bipolar Cautery, metal clip or Hem-o-lok clip will be used to seal the artery(ies)

SUMMARY:
Video assisted thoracoscopic surgery (VATS) anatomical lung resections (lobectomy or pneumonectomy) provide an effective minimally invasive treatment for stage 1 lung cancer.

Currently, a minority of anatomical pulmonary resections are being performed by VATS (15%) (6). The technical difficulty and danger of VATS lobectomy is related to pulmonary arterial branch manipulation and this is the main limitation of many thoracic surgeons regarding the adoption of VATS lobectomy. We believe that if we can decrease the manipulation required by the surgeon on the pulmonary arterial branch, we can make these procedures safe and therefore more prevalent for anatomical pulmonary resections.

DETAILED DESCRIPTION:
We believe that most of the stress (patient and surgeon) during VATS anatomical lung resection originates from manipulation of the pulmonary arteries. Endostaplers utilized during VATS to seal the pulmonary arteries require a lot of space and manipulation of these fragile vessels. Furthermore, the arteries must be completely dissected from the surrounding tissues. This increases manipulations of pulmonary arteries during the procedure. Energy sealing devices require much less space and dissection due to their size and sealing of the arteries can be performed without complete dissection from the surrounding tissues. Thus, the utilization of energy sealing devices will decrease excessive manipulations on the pulmonary arterial branches during VATS anatomical lung resections which can render these procedures easier and safer. This will not only decrease the stress on the patient, but also on the surgeon and will hopefully allow more surgeons to adopt these minimally invasive techniques which have been proven to be superior (length of stay, cost of care, pain, morbidity post-op, atrial fibrillation, quality of life, systemic inflammation, ability to receive adjuvant chemotherapy) to open thoracotomy.

The intraoperative techniques will not differ and blood vessel ligation will be performed according to standard operative procedures either using staplers or direct ligation of the pulmonary vessels.

After resection and delivery of the resected specimen out of the patient, the specimen will be examined in vitro out of the operative field in a non-sterile field in the operative room. The lobar pulmonary artery and its main segmental branches will be dissected. Canulation of a major segmental branch will be performed using an arterial pressure monitoring catheter. The canulation will be secured with ligation of 2-0 silk suture. A three way valve will be attached directly to the arterial catheter. One branch of the three way valve will be attached to a controlled pressure syringe pump and the other branch will be attached to a digital manometer. All other segmental branches of the pulmonary artery will be ligated to maintain the pressure throughout the catheterized segmental branch. Normal 25 mmHg pressure will be obtained by inflating with normal saline. The lobar pulmonary artery and the main segmental branches' diameters will be measured using a digital caliper from the adventitia to the adventitia in the inflated portion with normal saline of pressure 25 mmHg. The lobar pulmonary artery and the main segmental arteries will be sealed using one of the main energy seals (Ligasure, Harmonic scalpel, Enseal, Thunderbeat, unipolar or conventional bipolar cautery or application of metal or Hem-o-lok clips). The sealing will be performed with a normal 25 mmHg intra-arterial pressure.

In bipolar sealing, the arterial wall will be compressed between the energy device jaws until complete sealing is achieved. The artery will then be divided utilizing fine scissors. In pulmonary arterial branches sealed with Harmonic scalpel, Thunderbeat and Enseal, the arterial wall sealed will be divided in the same sealing step. In the Unipolar cautery arterial sealing, a DeBakey forceps will be utilized to compress the arterial walls together and then sealing will be performed with direct application of the unipolar cautery to the forceps. Complete sealing achieved by complete carbonization of the arterial walls. The artery will be divided with scissors after sealing.

After division of the pulmonary artery, normal saline solution will be injected through the controlled pressure syringe pump to achieve an intraluminal pressure until the bursting pressure is reached. Intraluminal pressure will be recorded and the bursting pressure will be registered.

The resected specimens will be divided into 8 groups according to the type of sealing performed; (Ligasure, Harmonic scalpel, Enseal, Thunderbeat, Unipolar and conventional bipolar cautery, Metal clip, and Hem-o-lok clip)

ELIGIBILITY:
Inclusion Criteria:

* All patients booked for open or VATS lobectomy, open or VATS pneumonectomy, lung transplantation.

Exclusion Criteria:

* Inability to consent for the study.
* Patients less than 18 years old.
* Hilar lung tumours with proximity to major pulmonary arteries that might affect the integrity of the vascular margin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome for analysis will be intergroup comparison of mean pulmonary artery burst pressures. | 1 month
  Intergroup differences will be compared with the student's t-test. Multivariable logistic regression models will be employed in order to compare burst pressures between groups controlling for potential confounder (disease state, size of vessel sealed, age of patient, pulmonary lobe…).

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Liberman M, Khereba M, Goudie E, Kazakov J, Thiffault V, Lafontaine E, Ferraro P. Pilot study of pulmonary arterial branch sealing using energy devices in an ex vivo model. J Thorac Cardiovasc Surg. 2014 Dec;148(6):3219-23. doi: 10.1016/j.jtcvs.2014.05.089. Epub 2014 Jul 19. PMID 25125207